CLINICAL TRIAL: NCT07085234
Title: The Efficacy and Safety of Iparomlimab/Tuvorlimab (QL1706) Combined With Modified TPF Regimen for Induction Therapy in Locally Advanced Nasopharyngeal Carcinoma
Brief Title: Iparomlimab/Tuvorlimab (QL1706) and Modified TPF Regimen for Induction Therapy in LANPC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Principal Investigator, San-Gang Wu, Clinical Professor, The First Affiliated Hospital of Xiamen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-113
Record Dates: First submitted 2025-06-30; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Locally Advanced Nasopharyngeal Carcinoma; Immunotherapy; Induction Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Iparomlimab/Tuvorlimab(QL-1706) and modified TPF regimen (Experimental): Patients will receive three cycles of Albumin-bound paclitaxel 260 mg/m² + cisplatin 75 mg/m² (divided on days 1 - 3) + S1 calculated according to body surface area, taken twice daily (days 1 - 14) + Iparomlimab/Tuvorlimab(QL-1706) 5 mg/kg (day 1).
  Interventions: Drug: Iparomlimab/Tuvorlimab(QL-1706) and modified TPF regimen

INTERVENTIONS:
Drug: Iparomlimab/Tuvorlimab(QL-1706) and modified TPF regimen — Induction therapy: Albumin-bound paclitaxel 260 mg/m² + cisplatin 75 mg/m² (divided on days 1 - 3) + S1 calculated according to body surface area, taken twice daily (days 1 - 14) + Iparomlimab/Tuvorlimab(QL-1706) 5 mg/kg (day 1). One cycle lasts for 21 days, and the treatment continues for three consecutive cycles.
  Concurrent chemotherapy: Cisplatin 80 mg/m², divided on days 1 - 3. One cycle lasts for 21 days, and the treatment continues for two consecutive cycles.
  Radiotherapy regimen: Whole-course IMRT.
  Other Names: QL-1706; Modified TPF regimen

SUMMARY:
This is a prospective, open-label, multicenter, single-arm clinical study. A total of 30 patients with locally advanced nasopharyngeal carcinoma who have not received prior systemic treatment are planned to be enrolled at three centers. After enrollment, the patients will receive induction therapy with Iparomlimab/Tuvorlimab(QL-1706) in combination with a modified TPF regimen, followed by concurrent chemoradiotherapy with cisplatin according to the standards of clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18 years old;
* Patients with nasopharyngeal carcinoma diagnosed by pathology (including histology or cytology), with a clinical stage of III - IV (excluding T3N0 - 1) (according to the UICC/AJCC TNM staging system (8th edition));
* No prior systematic treatment (surgery, radiotherapy, chemotherapy, etc.); At least one measurable lesion on imaging examination (according to RECIST criteria version 1.1);
* ECOG PS: 0 - 1 points;
* Expected survival time ≥ 3 months;
* Normal function of major organs, meeting the following criteria:

  1. Blood routine tests should meet the following (without blood transfusion within 14 days):

     1. HB ≥ 100 g/L,
     2. WBC ≥ 3 × 10⁹/L,
     3. ANC ≥ 1.5 × 10⁹/L,
     4. PLT ≥ 100 × 10⁹/L;
  2. Biochemical tests should meet the following criteria:

     1. BIL < 1.5 times the upper limit of normal (ULN),
     2. ALT and AST < 2.5 ULN, GPT ≤ 1.5 × ULN;
     3. Serum Cr ≤ 1 ULN, endogenous creatinine clearance rate > 60 ml/min (Cockcroft - Gault formula);
* Male subjects and women of childbearing potential must use contraception from the start of the first dose of the study drug until 24 weeks after the last dose of the study drug;
* Normal function of major organs, with basically normal blood routine, blood biochemistry and coagulation function tests;
* The investigator believes that the patient will benefit from the treatment in terms of survival;
* The patient voluntarily participates in this study and provides a written informed consent form.

Exclusion Criteria:

* Active, known, or suspected autoimmune diseases;
* Patients with hypertension whose blood pressure cannot be controlled within the normal range with antihypertensive medications (systolic blood pressure > 160 mmHg, diastolic blood pressure > 90 mmHg);
* Inherited bleeding tendency or coagulation disorders. Clinically significant bleeding symptoms occurred within 12 weeks before screening or there is a definite bleeding tendency (cumulative blood loss exceeding 50 ml within 24 hours);
* Uncontrolled cardiac clinical symptoms or diseases, such as: (1) Heart failure of NYHA class II or above; (2) Unstable angina; (3) Myocardial infarction within 24 weeks; (4) Clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention;
* Interstitial lung disease, drug-induced pneumonia, radiation pneumonia requiring steroid treatment, active pneumonia with clinical symptoms, or severe pulmonary function impairment;
* Subjects with active hepatitis B (HBV DNA ≥ 2000 IU/mL or 10⁴ copies/mL) or hepatitis C (positive for hepatitis C antibody and HCV-RNA above the lower limit of detection of the analytical method);
* Subjects with allergic reactions to the drugs used in this study;
* Pregnant or lactating women;
* Other conditions considered by the investigator as unsuitable for participation in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete response rates after induction therapy | From the time of enrollment to the end of cycle 3 of induction therapy (each cycle is 21 days).
  Higher scores mean a better outcome.

SECONDARY OUTCOMES:
ORR | From the time of enrollment to the end of cycle 3 of induction therapy (each cycle is 21 days).
  Higher scores mean a better outcome.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | From the time of enrollment to the end of cycle 3 of induction therapy (each cycle is 21 days).
  Higher scores mean a worse outcome.
PFS | From the time of enrollment until two years after the completion of the treatment.
  Higher scores mean a better outcome.
OS | From the time of enrollment until two years after the completion of the treatment
  Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No